CLINICAL TRIAL: NCT07287943
Title: Efficacy and Safety of Medtronic 780G Automated Insulin Delivery System in Adults With Type 1 Diabetes and Gastroparesis
Brief Title: To Study the Efficacy and Safety of Medtronic 780G Insulin Pump in People With Gastroparesis and Type 1 Diabetes.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Viral N. Shah (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor-Investigator, Viral N. Shah, Principal Investigator, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 28244
Record Dates: First submitted 2025-12-14; First posted 2025-12-17 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Type 1 Diabetes; Gastroparesis Due to Diabetes Mellitus Type I
Keywords: type 1 diabetes; gastroparesis
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Gastroparesis | interventions — Insemination, Artificial, Heterologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Medtronic 780G group (Experimental)
  Interventions: Device: Medtronic 780G AID
- Usual care (No Intervention): Participants will continue either multiple daily injections or other insulin pumps in non automated mode

INTERVENTIONS:
Device: Medtronic 780G AID — Participants in Medtronic AID treatment group will use it for three months
  Arms: Medtronic 780G group

SUMMARY:
The goal of this clinical trial is to learn if Medtronic 780G automated insulin delivery system improves high blood sugars in adult persons with type 1 diabetes and gastroparesis. It will also learn about the safety of this system. Main questions it aims to answer are:

Does Medtronic 780G automated insulin delivery system (insulin pump) improve blood glucose in range from start of study to 3months.

Researchers will compare Medtronic 780G automated insulin delivery system with usual care (multiple daily insulin injection use or other insulin pumps) to see if it improves blood glucose.

Participants will:

Use Medtronic 780G automated insulin delivery system or continue with usual care for 3 months.

Visit the clinic in person (3 visits) or via phone (four visits) over 3 months for review of blood glucose readings and follow up of symptoms.

Ingest a special meal to see how it affects blood sugars (optional)

It is expected that a total of up to 34 person with type 1 diabetes and gastroparesis will be recruited through adult outpatient diabetes and gastroenterology clinics of the investigation centre.

DETAILED DESCRIPTION:
STUDY OBJECTIVE To evaluate efficacy (change in time spent in 70-180 mg/dL, TIR) and safety of Medtronic 780 G compared to usual care in adults with T1D and gastroparesis.

OUTCOMES

Primary outcome Time spent in sensor glucose of 70-180 mg/dL

Secondary outcomes

1. HbA1c
2. Mean glucose
3. Percent time spent in sensor glucose range of 70-140 mg/dL (time in tight target range; TTIR)
4. Percent time spent in sensor glucose >180 mg/dL and >250 mg/dL
5. Percent time spent in sensor glucose<70 mg/dL and <54 mg/dL
6. Glucose variability (standard deviation (SD) of glucose)

Safety Outcomes:

1. Severe hypoglycemia (SH)
2. Diabetic ketoacidosis (DKA)

Exploratory Outcomes

1. Proportion of patients achieving HbA1c <7%
2. Proportion of patients achieving TIR >70%
3. Proportion of patients achieving HbA1c <7.5%
4. Proportion of patients achieving TITR >55%
5. Primary and secondary outcomes by bolusing/day (no bolus or 1 per day vs at least 2 boluses/day)
6. Patient reported outcomes (PRO): device satisfaction, diabetes distress, PAGI-SYM (Patient assessment of GI Symptoms) score, GCSI (Gastroparesis Cardinal Symptom Index) and PAGI-QOL (Quality of Life) score

STUDY DESIGN

This will a prospective, open label, randomized clinical trial with 1:1 randomization to an intervention group using the study Medtronic 780G AID system versus usual care (either multiple daily injections (MDI) or insulin pump along with continuous glucose monitoring (CGM) for 12 weeks.

STUDY POPULATION Inclusion criteria

1. Age ≥18 years
2. Diagnosis of T1D for at least 12 months with stable insulin regimen for at least 2 months
3. HbA1c ≥8.0%
4. Diagnosis of gastroparesis per National Institute of Health (NIH) definition for at least 2 years.
5. Willing to use Medtronic 780G system either with Guardian Connect 4 or Simplera CGM.
6. Ability to provide informed consent before any trial-related activities
7. If randomized to usual care group and on an insulin pump already, should be willing to use pump in manual mode only for the duration of the study

Exclusion criteria

1. Age <18 years
2. Current use of inhaled insulin (Afrezza)
3. Patients with T1D using any glucose lowering medications other than insulin at the time of screening
4. Pregnancy, breast feeding, or wanting to become pregnant
5. Current use (≥ 2 weeks of continuous use) of any steroidal medication, or anticipated long-term steroidal treatment (>4 weeks continuously), during the study period
6. History of gastric outlet obstruction or other gastrointestinal structural abnormalities
7. Estimated glomerular filtration rate (eGFR) <30 or on dialysis
8. History of SH in the previous 3 months
9. History of two or more episodes DKA requiring hospitalization in the past 12 months
10. Any medical (such as severe cardiovascular disease, malignancy, chronic liver disease) or psychosocial conditions that make a person unfit for the study at the discretion of investigators
11. Use of investigational drugs within 5 half-lives prior to screening
12. Current use of cannabis or history of cannabinoid hyperemesis syndrome Withdrawal criteria

    * Participation in this research is voluntary. Subjects may withdraw at will at any time. When withdrawing from the study, the participant should let the research team know that he/she wishes to withdraw. A participant may provide the research team with the reason(s) for leaving the study but is not required to provide their reason.
    * Participants will be withdrawn from the study if they become pregnant, actively try to become pregnant or at the judgement of investigators due to safety concerns.
    * After withdrawal, the participant will be given instructions on how to correctly and safely return to the previous treatment regimen. Instructions are also given on who to contact if there are any questions or concerns that arise after study withdrawal.
    * At the time of withdrawal, the research participant should let the research team know if he/she will allow the use of his/her health information and collected data by the researchers.

    Subject replacement Withdrawn subjects will not be replaced. However, re-screening is allowed within recruitment period at the investigator's discretion.

    Reminders To minimize loss to follow-up, reminders (text message, phone call or email) will be sent to participants prior to each clinic visits.

    VISIT PROCEDURES:
    * In brief, there are up to three in-person research visits and up to four phone call visits.

      * Before screening takes place, subjects will be provided with written information about the trial and the procedures involved. Subjects will be fully informed, both orally and in writing, about their responsibilities and rights while participating in the trial, as well as about possible advantages and disadvantages when participating in this trial. Subjects will have the opportunity to ask questions and have ample time to consider participation. The informed consent process will take place before the screening visit. Before signing the informed consent, the investigator will make sure that the potential subject has full knowledge of the study processes, and the possibility to withdrawal at any time during the study.
      * Subjects who wish to enroll in the trial must sign and date the informed consent form for the trial before participating in any trial-related procedures. All subjects will be provided with a copy of signed informed consent form.

    Screening (Visit 1 in-person)

    • The subjects will be assigned a unique subject number, which will remain the same throughout the trial. The subject number will consist of 2 digits (e.g. 01).
    * All subjects will undergo review of inclusion and exclusion criteria.
    * Medical history, concomitant medications and demographics data will be recorded.
    * Patients will be told the importance of compliance of the pre-set study visit time schedules.
    * All subjects will be assessed and reeducated on diabetes self-management, appropriate and safe use of their own diabetes devices, and its trouble shooting, prevention and treatment of hypoglycemia and sick day management.
    * All subjects must use appropriate insulin that is approved for their hybrid closed loop system.
    * A blinded CGM will be provided to all participants to be used for 14 days.
    * Point of care (POC) A1c will be obtained for screening.
    * PAGI-SYM (Patient assessment of GI Symptoms) score, GCSI (Gastroparesis Cardinal Symptom Index), PAGI-QOL (Quality of Life) score will be administered.
    * All participants will be given the option of ingesting standardized meal traditionally used to evaluate gastric emptying. Participants will pick a day between day 2 to day 6 of CGM wear, to ingest this at home after 8 hours of fasting, followed by nothing per mouth except water for next 4 hours.

    Reminder Call 1

    • Participants who agreed to ingest gastric emptying study test meal will be reminded by the study coordinator one day prior to at home test meal ingestion (details in Procedure manual). The study coordinator will also go over the instruction leaflet.

    Randomization (Visit 2 in-person)
    * Randomization visit will be done within 2 weeks from screening visit.
    * Subjects who use the blinded CGM for at least 7 days will be randomized. The rest will be offered a screening extension and will receive randomization accordingly.
    * Subjects will be randomized using computer generated randomization scheme to receive either using the study Medtronic 780G AID system versus usual care, either MDI or personal insulin pump along with CGM for 12 weeks.
    * Pump Training for Medtronic 780G AID system will be conducted for those randomized to Medtronic 780 G group.
    * A blinded CGM will be provided to those participants in usual care group who are using their personal CGM to be used for 14 days.
    * Those who will be randomized to usual care and are CGM naïve will be provided Medtronic GC 4 or Simplera for the study duration.
    * Medical history and medications will be reviewed for any changes.
    * A1c via Central Lab

    Reminder Call 2 (only for intervention group) • Intervention group will be reminded on day 2 to turn on their Smart Guard system.

    Phone visit 1
    * This will occur at 7±2 days of randomization.
    * Insulin delivery and CGM data will be reviewed for insulin dose adjustment and/or pump settings.
    * AE assessment Phone visit 2
    * This will occur at 14±3 days of randomization.
    * Medical history and medications will be reviewed for any changes.
    * Insulin delivery and CGM data will be reviewed for insulin dose adjustment and/or pump settings.
    * AE assessment . Phone visit 3
    * This will occur at 30±3 days of randomization.
    * Medical history and medications will be reviewed for any changes.
    * Insulin delivery and CGM data will be reviewed for insulin dose adjustment and/or pump settings.
    * AE assessment Phone visit 4
    * This will occur after 60±3 days of randomization.
    * Medical history and medications will be reviewed for any changes.
    * Insulin delivery and CGM data will be reviewed for insulin dose adjustment and/or pump settings.
    * AE assessment

    Reminder Call 3

    • Participants in usual care group who are using their personal CGM will be reminded to self-apply blinded CGM two weeks prior to last in person visit.

    Visit 3 in-person

    • This will occur after 90±7 days of randomization.

    • Medical history and medications will be reviewed for any changes.

    • Insulin delivery and CGM data will be reviewed for insulin dose adjustment and/or pump settings.

    • AE assessment

    • PAGI-SYM (Patient assessment of GI Symptoms) score, GCSI (Gastroparesis Cardinal Symptom Index), PAGI-QOL (Quality of Life) score will be administered.
    * A1c via Central Lab

      * STATISTICAL PLAN Sample size calculation Based on prior studies of CGM-based interventions in adults with T1D, we estimate the standard deviation (SD) of TIR to be approximately 10.4%. We aim to detect a clinically meaningful difference of 10 percentage points in change from baseline (delta) TIR between the intervention group (Medtronic 780G system) and the control group (usual care), with a two-sided alpha of 0.05 and 80% power. Using a two-sample t-test (appropriate due to small sample size and unknown population SD), the required sample size per group is 17 participants, totaling 34 completers. To allow for a 15% dropout rate, we will randomize 40 participants (20 per group).

    Analysis Plan

    Primary Outcome The primary efficacy endpoint is the change in percentage of time in range (TIR; sensor glucose 70-180 mg/dL) from baseline to 3 months. The main comparison focuses on the between-group difference in this change from baseline (time in range calculated using 2 weeks of CGM data prior to randomization) to 3 month (2 weeks of CGM prior to Week 12). An independent two-sample t-test (or Mann-Whitney U test if normality assumptions are violated) will be used to compare the primary outcome between groups.

    Given the availability of CGM data at multiple timepoints, linear mixed-effects models (LMMs) will be used to analyze changes in TIR over time. These models will include random intercepts for participants (to account for within-subject correlation) and fixed effects for time, treatment group, and their interaction. This approach will assess both overall treatment effects and time-by-treatment interactions.

    Secondary Outcomes

    Secondary outcomes will be analyzed using a similar statistical framework as the primary outcome. Specifically, changes from baseline to 3 months in each secondary endpoint will be compared between the two randomized groups (Medtronic 780G vs usual care) using independent two-sample t-tests (or non-parametric alternatives, such as the Mann-Whitney U test, when assumptions of normality are violated). Where appropriate, analysis of covariance (ANCOVA) models will be used to adjust for baseline values and improve precision.

    Safety Outcomes Severe hypoglycemia and DKA events will be compared between two groups. We will calculate events (%) and number of participants with the event between two groups. We will also populate adverse events between two groups. No formal statistical analysis will be conducted for adverse events between two groups given that SH and DKA events are rare and small sample size of the study.

    Missing Data Handling CGM Data Completeness: CGM data quality will be assessed for each 14-day wear period. For descriptive purposes, a threshold of ≥50% CGM wear time (equivalent to ≥7 full days of data) will be used to characterize data completeness.

    Approach to Missing Outcome Data: All randomized participants will be included in the analysis under the ITT framework. For missing CGM outcome data, we will use appropriate statistical techniques such as multiple imputation or maximum likelihood estimation, assuming that data are missing at random (MAR).

    Statistical Significance and Interpretation

    • All hypothesis tests will be two-tailed with a significance level (α) set at 0.05.

    • For secondary and exploratory outcomes involving multiple comparisons, false discovery rate (FDR) will be controlled using the Benjamini-Hochberg procedure to reduce the risk of type I error.

    • 95% confidence intervals (CIs) will be reported for all point estimates to convey the precision and clinical relevance of findings, regardless of statistical significance.

    • Effect sizes (e.g., mean differences, standardized effect sizes) will be reported where appropriate to aid interpretation beyond p-values.

    STUDY DEVICES AND MATERIALS • Patients will be using their own insulin in both groups.

    • At screening all participants will receive blinded CGM for 14 days.
    * Participants randomized to 780 G will receive pump and CGM supplies for the duration of the trial.
    * Participants randomized to usual care will be using their own insulin delivery methods
    * Those who are naïve to CGM, will be provided with CGM (either Medtronic GC4 or Simplera) throughout the trial.
    * Participants in usual care group who will use personal CGM will receive blinded CGM at two different time points: randomization and 2 weeks prior to last in-person visit.

ELIGIBILITY:
Inclusion Criteria:

* 5. STUDY POPULATION 5.1 Inclusion criteria
* Age ≥18 years
* Diagnosis of T1D for at least 12 months with stable insulin regimen for at least 2 months
* HbA1c ≥8.0%
* Diagnosis of gastroparesis per National Institute of Health (NIH) definition for at least 2 years.
* Willing to use Medtronic 780G system either with Guardian Connect 4 or Simplera CGM.
* Ability to provide informed consent before any trial-related activities
* If randomized to usual care group and on an insulin pump already, should be willing to use pump in manual mode only for the duration of the study

5.2 Exclusion criteria

* Age <18 years
* Current use of inhaled insulin (Afrezza)
* Patients with T1D using any glucose lowering medications other than insulin at the time of screening
* Pregnancy, breast feeding, or wanting to become pregnant
* Current use (≥ 2 weeks of continuous use) of any steroidal medication, or anticipated long-term steroidal treatment (>4 weeks continuously), during the study period
* History of gastric outlet obstruction or other gastrointestinal structural abnormalities
* Estimated glomerular filtration rate (eGFR) <30 or on dialysis
* History of SH in the previous 3 months
* History of two or more episodes DKA requiring hospitalization in the past 12 months
* Any medical (such as severe cardiovascular disease, malignancy, chronic liver disease) or psychosocial conditions that make a person unfit for the study at the discretion of investigators
* Use of investigational drugs within 5 half-lives prior to screening
* Current use of cannabis or history of cannabinoid hyperemesis syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the change in percentage of time in range (TIR; sensor glucose 70-180 mg/dL) from baseline to 3 months. The main comparison focuses on the between-group difference in this change from baseline. | 3months

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Health, Univeristy hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
not for now